CLINICAL TRIAL: NCT05234177
Title: Tempus CRC Surveillance Study: A Longitudinal Circulating Tumor DNA (ctDNA) Biomarker Profiling Study of Patients With Colorectal Cancer (CRC) Using Comprehensive Next-Generation Sequencing (NGS)Assays
Brief Title: Tempus CRC Surveillance Study: A ctDNA Biomarker Profiling Study of Patients With CRC Using NGS Assays
Status: Recruiting | Type: Observational
Sponsor: Tempus AI (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CA-004
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: Cancer; Oncology; Observational; Genomic Profiling; Precision medicine; CRC; Colorectal Cancer; NGS; Biomarkers
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with stage I-IV colorectal cancer (CRC): This protocol will include participants with stage I-IV CRC who are scheduled to undergo or have undergone a surgical resection with curative intent.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention

SUMMARY:
The study is an observational multicenter evaluation of participants with colorectal cancer (CRC) who will receive longitudinal plasma ctDNA biomarker profiling in addition to their standard-of-care therapy and disease surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected colorectal adenocarcinoma (Stage I to IVA disease)
* Planning to undergo or has undergone a surgical resection for suspected adenocarcinoma of the colon or rectum with curative intent.
* 18 years old or older
* Willing and able to provide informed consent
* Willing to have additional blood samples collected during routine surveillance visits

Exclusion Criteria:

* Not willing to have additional blood samples collected
* Pathology that is not consistent with colorectal adenocarcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This protocol targets patients with colorectal cancer (CRC), stage I-IVA disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival | 2 years
  Recurrence-Free Survival as assessed by standard radiographic imaging, measured from the day of completion of definitive treatment to first radiographic recurrence or death

SECONDARY OUTCOMES:
Sensitivity | 2 years
  Sensitivity defined as the proportion of participants who develop recurrence who have ctDNA detected.
Specificity | 2 years
  Specificity defined as the proportion of participants who do not develop recurrence who do not have ctDNA detected.
Positive Predictive Value | 2 years
  Positive predictive value (PPV) defined as the proportion of participants who have ctDNA detected who recur.

OTHER OUTCOMES:
Overall Survival | 2 years or until the patient is reported deceased
  The duration of time between enrollment and death for any reason
Lead Time | 2 years
  Lead time defined as the interval between ctDNA detection and clinical detection of recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Kristiyana Kaneva, MD, MS, Principal Investigator — Tempus AI, Inc.
Locations (20):
- United States (20):
  - Mercy Clinic Oncology - Fort Smith, Fort Smith, Arkansas
  - MemorialCare, Fountain Valley, California
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Mercy Clinic Oncology and Hematology - Joplin, Joplin, Missouri
  - Mercy Clinic Cancer and Hematology - Chub O'Reilly Cancer Center, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Clinic Oncology and Hematology - Sindelar Cancer Center, St Louis, Missouri
  - Mercy Clinic Oncology and Hematology - David C. Pratt Cancer Center, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Aultman Hospital, Canton, Ohio
  - TriHealth Cancer Institute, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Mercy Clinic Oncology and Hematology - Coletta, Oklahoma City, Oklahoma
  - Cancer Care Associates of York, York, Pennsylvania
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Washington / Fred Hutchinson Cancer Center, Seattle, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] Siegel RL, Miller KD, Goding Sauer A, Fedewa SA, Butterly LF, Anderson JC, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2020. CA Cancer J Clin. 2020 May;70(3):145-164. doi: 10.3322/caac.21601. Epub 2020 Mar 5. PMID 32133645
- [Background] Stoffel EM, Murphy CC. Epidemiology and Mechanisms of the Increasing Incidence of Colon and Rectal Cancers in Young Adults. Gastroenterology. 2020 Jan;158(2):341-353. doi: 10.1053/j.gastro.2019.07.055. Epub 2019 Aug 5. PMID 31394082
- [Background] Islami F, Ward EM, Sung H, Cronin KA, Tangka FKL, Sherman RL, Zhao J, Anderson RN, Henley SJ, Yabroff KR, Jemal A, Benard VB. Annual Report to the Nation on the Status of Cancer, Part 1: National Cancer Statistics. J Natl Cancer Inst. 2021 Nov 29;113(12):1648-1669. doi: 10.1093/jnci/djab131. PMID 34240195
- [Background] Brenner H, Kloor M, Pox CP. Colorectal cancer. Lancet. 2014 Apr 26;383(9927):1490-1502. doi: 10.1016/S0140-6736(13)61649-9. Epub 2013 Nov 11. PMID 24225001
- [Background] Institute NC, National Cancer Institute. AJCC Cancer Staging Manual 8th Edition. Definitions. 2020
- [Background] Leufkens AM, van den Bosch MA, van Leeuwen MS, Siersema PD. Diagnostic accuracy of computed tomography for colon cancer staging: a systematic review. Scand J Gastroenterol. 2011 Jul;46(7-8):887-94. doi: 10.3109/00365521.2011.574732. Epub 2011 Apr 20. PMID 21504379
- [Background] Benson AB 3rd, Choti MA, Cohen AM, Doroshow JH, Fuchs C, Kiel K, Martin EW Jr, McGinn C, Petrelli NJ, Posey JA, Skibber JM, Venook A, Yeatman TJ; National Comprehensive Cancer Network. NCCN Practice Guidelines for Colorectal Cancer. Oncology (Williston Park). 2000 Nov;14(11A):203-12. PMID 11195411
- [Background] Kahi CJ, Boland CR, Dominitz JA, Giardiello FM, Johnson DA, Kaltenbach T, Lieberman D, Levin TR, Robertson DJ, Rex DK; United States Multi-Society Task Force on Colorectal Cancer. Colonoscopy Surveillance After Colorectal Cancer Resection: Recommendations of the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2016 Mar;150(3):758-768.e11. doi: 10.1053/j.gastro.2016.01.001. Epub 2016 Feb 10. PMID 26892199
- [Background] Winawer SJ, Fletcher RH, Miller L, Godlee F, Stolar MH, Mulrow CD, Woolf SH, Glick SN, Ganiats TG, Bond JH, Rosen L, Zapka JG, Olsen SJ, Giardiello FM, Sisk JE, Van Antwerp R, Brown-Davis C, Marciniak DA, Mayer RJ. Colorectal cancer screening: clinical guidelines and rationale. Gastroenterology. 1997 Feb;112(2):594-642. doi: 10.1053/gast.1997.v112.agast970594. No abstract available. PMID 9024315
- [Background] Provenzale D, Ness RM, Llor X, Weiss JM, Abbadessa B, Cooper G, Early DS, Friedman M, Giardiello FM, Glaser K, Gurudu S, Halverson AL, Issaka R, Jain R, Kanth P, Kidambi T, Lazenby AJ, Maguire L, Markowitz AJ, May FP, Mayer RJ, Mehta S, Patel S, Peter S, Stanich PP, Terdiman J, Keller J, Dwyer MA, Ogba N. NCCN Guidelines Insights: Colorectal Cancer Screening, Version 2.2020. J Natl Compr Canc Netw. 2020 Oct 1;18(10):1312-1320. doi: 10.6004/jnccn.2020.0048. PMID 33022639
- [Background] Ladabaum U, Dominitz JA, Kahi C, Schoen RE. Strategies for Colorectal Cancer Screening. Gastroenterology. 2020 Jan;158(2):418-432. doi: 10.1053/j.gastro.2019.06.043. Epub 2019 Aug 5. PMID 31394083
- [Background] Muller MF, Ibrahim AE, Arends MJ. Molecular pathological classification of colorectal cancer. Virchows Arch. 2016 Aug;469(2):125-34. doi: 10.1007/s00428-016-1956-3. Epub 2016 Jun 20. PMID 27325016
- [Background] Poulogiannis G, Ichimura K, Hamoudi RA, Luo F, Leung SY, Yuen ST, Harrison DJ, Wyllie AH, Arends MJ. Prognostic relevance of DNA copy number changes in colorectal cancer. J Pathol. 2010 Feb;220(3):338-47. doi: 10.1002/path.2640. PMID 19911421
- [Background] Arends MJ. Pathways of colorectal carcinogenesis. Appl Immunohistochem Mol Morphol. 2013 Mar;21(2):97-102. doi: 10.1097/PAI.0b013e31827ea79e. PMID 23417071
- [Background] Poulogiannis G, Frayling IM, Arends MJ. DNA mismatch repair deficiency in sporadic colorectal cancer and Lynch syndrome. Histopathology. 2010 Jan;56(2):167-79. doi: 10.1111/j.1365-2559.2009.03392.x. PMID 20102395
- [Background] Giardiello FM, Allen JI, Axilbund JE, Boland CR, Burke CA, Burt RW, Church JM, Dominitz JA, Johnson DA, Kaltenbach T, Levin TR, Lieberman DA, Robertson DJ, Syngal S, Rex DK. Guidelines on genetic evaluation and management of Lynch syndrome: a consensus statement by the US Multi-Society Task Force on Colorectal Cancer. Dis Colon Rectum. 2014 Aug;57(8):1025-48. doi: 10.1097/DCR.000000000000000. PMID 25003300
- [Background] Domingo E, Niessen RC, Oliveira C, Alhopuro P, Moutinho C, Espin E, Armengol M, Sijmons RH, Kleibeuker JH, Seruca R, Aaltonen LA, Imai K, Yamamoto H, Schwartz S Jr, Hofstra RM. BRAF-V600E is not involved in the colorectal tumorigenesis of HNPCC in patients with functional MLH1 and MSH2 genes. Oncogene. 2005 Jun 2;24(24):3995-8. doi: 10.1038/sj.onc.1208569. PMID 15782118
- [Background] Morse MA, Hochster H, Benson A. Perspectives on Treatment of Metastatic Colorectal Cancer with Immune Checkpoint Inhibitor Therapy. Oncologist. 2020 Jan;25(1):33-45. doi: 10.1634/theoncologist.2019-0176. Epub 2019 Aug 5. PMID 31383813
- [Background] Overman MJ, McDermott R, Leach JL, Lonardi S, Lenz HJ, Morse MA, Desai J, Hill A, Axelson M, Moss RA, Goldberg MV, Cao ZA, Ledeine JM, Maglinte GA, Kopetz S, Andre T. Nivolumab in patients with metastatic DNA mismatch repair-deficient or microsatellite instability-high colorectal cancer (CheckMate 142): an open-label, multicentre, phase 2 study. Lancet Oncol. 2017 Sep;18(9):1182-1191. doi: 10.1016/S1470-2045(17)30422-9. Epub 2017 Jul 19. PMID 28734759
- [Background] Rotte A. Combination of CTLA-4 and PD-1 blockers for treatment of cancer. J Exp Clin Cancer Res. 2019 Jun 13;38(1):255. doi: 10.1186/s13046-019-1259-z. PMID 31196207
- [Background] Gourd E. Nivolumab plus ipilimumab in metastatic colorectal cancer. Lancet Oncol. 2018 Mar;19(3):e139. doi: 10.1016/S1470-2045(18)30067-6. Epub 2018 Jan 26. No abstract available. PMID 29395861
- [Background] Overman MJ, Lonardi S, Wong KYM, Lenz HJ, Gelsomino F, Aglietta M, Morse MA, Van Cutsem E, McDermott R, Hill A, Sawyer MB, Hendlisz A, Neyns B, Svrcek M, Moss RA, Ledeine JM, Cao ZA, Kamble S, Kopetz S, Andre T. Durable Clinical Benefit With Nivolumab Plus Ipilimumab in DNA Mismatch Repair-Deficient/Microsatellite Instability-High Metastatic Colorectal Cancer. J Clin Oncol. 2018 Mar 10;36(8):773-779. doi: 10.1200/JCO.2017.76.9901. Epub 2018 Jan 20. PMID 29355075
- [Background] Noffsinger AE. Serrated polyps and colorectal cancer: new pathway to malignancy. Annu Rev Pathol. 2009;4:343-64. doi: 10.1146/annurev.pathol.4.110807.092317. PMID 19400693
- [Background] Kopetz S, Grothey A, Yaeger R, Van Cutsem E, Desai J, Yoshino T, Wasan H, Ciardiello F, Loupakis F, Hong YS, Steeghs N, Guren TK, Arkenau HT, Garcia-Alfonso P, Pfeiffer P, Orlov S, Lonardi S, Elez E, Kim TW, Schellens JHM, Guo C, Krishnan A, Dekervel J, Morris V, Calvo Ferrandiz A, Tarpgaard LS, Braun M, Gollerkeri A, Keir C, Maharry K, Pickard M, Christy-Bittel J, Anderson L, Sandor V, Tabernero J. Encorafenib, Binimetinib, and Cetuximab in BRAF V600E-Mutated Colorectal Cancer. N Engl J Med. 2019 Oct 24;381(17):1632-1643. doi: 10.1056/NEJMoa1908075. Epub 2019 Sep 30. PMID 31566309
- [Background] Lievre A, Bachet JB, Boige V, Cayre A, Le Corre D, Buc E, Ychou M, Bouche O, Landi B, Louvet C, Andre T, Bibeau F, Diebold MD, Rougier P, Ducreux M, Tomasic G, Emile JF, Penault-Llorca F, Laurent-Puig P. KRAS mutations as an independent prognostic factor in patients with advanced colorectal cancer treated with cetuximab. J Clin Oncol. 2008 Jan 20;26(3):374-9. doi: 10.1200/JCO.2007.12.5906. PMID 18202412
- [Background] Douillard JY, Oliner KS, Siena S, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Williams R, Rong A, Wiezorek J, Sidhu R, Patterson SD. Panitumumab-FOLFOX4 treatment and RAS mutations in colorectal cancer. N Engl J Med. 2013 Sep 12;369(11):1023-34. doi: 10.1056/NEJMoa1305275. PMID 24024839
- [Background] Lai E, Liscia N, Donisi C, Mariani S, Tolu S, Pretta A, Persano M, Pinna G, Balconi F, Pireddu A, Impera V, Dubois M, Migliari M, Spanu D, Saba G, Camera S, Musio F, Ziranu P, Puzzoni M, Demurtas L, Pusceddu V, Dettori M, Massa E, Atzori F, Dessi M, Astara G, Madeddu C, Scartozzi M. Molecular-Biology-Driven Treatment for Metastatic Colorectal Cancer. Cancers (Basel). 2020 May 13;12(5):1214. doi: 10.3390/cancers12051214. PMID 32413973
- [Background] Normanno N, Cervantes A, Ciardiello F, De Luca A, Pinto C. The liquid biopsy in the management of colorectal cancer patients: Current applications and future scenarios. Cancer Treat Rev. 2018 Nov;70:1-8. doi: 10.1016/j.ctrv.2018.07.007. Epub 2018 Jul 18. PMID 30053724
- [Background] Siravegna G, Marsoni S, Siena S, Bardelli A. Integrating liquid biopsies into the management of cancer. Nat Rev Clin Oncol. 2017 Sep;14(9):531-548. doi: 10.1038/nrclinonc.2017.14. Epub 2017 Mar 2. PMID 28252003
- [Background] Crowley E, Di Nicolantonio F, Loupakis F, Bardelli A. Liquid biopsy: monitoring cancer-genetics in the blood. Nat Rev Clin Oncol. 2013 Aug;10(8):472-84. doi: 10.1038/nrclinonc.2013.110. Epub 2013 Jul 9. PMID 23836314
- [Background] Kolencik D, Shishido SN, Pitule P, Mason J, Hicks J, Kuhn P. Liquid Biopsy in Colorectal Carcinoma: Clinical Applications and Challenges. Cancers (Basel). 2020 May 27;12(6):1376. doi: 10.3390/cancers12061376. PMID 32471160
- [Background] Richman SD, Chambers P, Seymour MT, Daly C, Grant S, Hemmings G, Quirke P. Intra-tumoral heterogeneity of KRAS and BRAF mutation status in patients with advanced colorectal cancer (aCRC) and cost-effectiveness of multiple sample testing. Anal Cell Pathol (Amst). 2011;34(1-2):61-6. doi: 10.3233/ACP-2011-0005. PMID 21483104
- [Background] Kasi PM, Sawyer S, Guilford J, Munro M, Ellers S, Wulff J, Hook N, Krinshpun S, Koyen Malashevich A, Malhotra M, Rodriguez A, Moshkevich S, Grothey A, Kopetz S, Billings P, Aleshin A. BESPOKE study protocol: a multicentre, prospective observational study to evaluate the impact of circulating tumour DNA guided therapy on patients with colorectal cancer. BMJ Open. 2021 Sep 24;11(9):e047831. doi: 10.1136/bmjopen-2020-047831. PMID 34561256
- [Background] Hu Y, Ulrich BC, Supplee J, Kuang Y, Lizotte PH, Feeney NB, Guibert NM, Awad MM, Wong KK, Janne PA, Paweletz CP, Oxnard GR. False-Positive Plasma Genotyping Due to Clonal Hematopoiesis. Clin Cancer Res. 2018 Sep 15;24(18):4437-4443. doi: 10.1158/1078-0432.CCR-18-0143. Epub 2018 Mar 22. PMID 29567812
- [Background] Parikh AR, Van Seventer EE, Siravegna G, Hartwig AV, Jaimovich A, He Y, Kanter K, Fish MG, Fosbenner KD, Miao B, Phillips S, Carmichael JH, Sharma N, Jarnagin J, Baiev I, Shah YS, Fetter IJ, Shahzade HA, Allen JN, Blaszkowsky LS, Clark JW, Dubois JS, Franses JW, Giantonio BJ, Goyal L, Klempner SJ, Nipp RD, Roeland EJ, Ryan DP, Weekes CD, Wo JY, Hong TS, Bordeianou L, Ferrone CR, Qadan M, Kunitake H, Berger D, Ricciardi R, Cusack JC, Raymond VM, Talasaz A, Boland GM, Corcoran RB. Minimal Residual Disease Detection using a Plasma-only Circulating Tumor DNA Assay in Patients with Colorectal Cancer. Clin Cancer Res. 2021 Oct 15;27(20):5586-5594. doi: 10.1158/1078-0432.CCR-21-0410. Epub 2021 Apr 29. PMID 33926918
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Beaubier N, Bontrager M, Huether R, Igartua C, Lau D, Tell R, Bobe AM, Bush S, Chang AL, Hoskinson DC, Khan AA, Kudalkar E, Leibowitz BD, Lozachmeur A, Michuda J, Parsons J, Perera JF, Salahudeen A, Shah KP, Taxter T, Zhu W, White KP. Integrated genomic profiling expands clinical options for patients with cancer. Nat Biotechnol. 2019 Nov;37(11):1351-1360. doi: 10.1038/s41587-019-0259-z. Epub 2019 Sep 30. PMID 31570899
- [Background] Beaubier N, Tell R, Lau D, Parsons JR, Bush S, Perera J, Sorrells S, Baker T, Chang A, Michuda J, Iguartua C, MacNeil S, Shah K, Ellis P, Yeatts K, Mahon B, Taxter T, Bontrager M, Khan A, Huether R, Lefkofsky E, White KP. Clinical validation of the tempus xT next-generation targeted oncology sequencing assay. Oncotarget. 2019 Mar 22;10(24):2384-2396. doi: 10.18632/oncotarget.26797. eCollection 2019 Mar 22. PMID 31040929